CLINICAL TRIAL: NCT03534388
Title: A Feasibility Study to Evaluate a Skin Cleansing Regimen With a Sodium Hypochlorite Wash in Lower Extremity Arterial Bypass Graft Surgery or Femoral Endarterectomy
Brief Title: A Feasibility Study to Evaluate Skin Cleansing With a Sodium Hypochlorite Wash
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulty
Sponsor: TopMD Skin Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLN 004.2
Record Dates: First submitted 2017-11-30; First posted 2018-05-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2018-05

CONDITIONS: Arterial Bypass Graft Surgery

STUDY DESIGN:
Intervention Model Description: Feasibility comparing to retrospective data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Subjects (Other)
  Interventions: Other: Sodium Hypochlorite Cleanser

INTERVENTIONS:
Other: Sodium Hypochlorite Cleanser — Cleansing with CLn BodyWash

SUMMARY:
Feasibility study in approximately 20 subjects to investigate the rate of infection with subjects undergoing elective lower extremity arterial bypass graft surgery or femoral endarterectomy. The subjects are instructed to shower with the sodium hypochlorite body wash daily, or as modified by the physician, for 5 of the 7 days leading to their surgery.

DETAILED DESCRIPTION:
This is a feasibility study in approximately 20 subjects over a 5-week period per subject. The study will investigate the rate of infection with subjects undergoing elective lower extremity arterial bypass graft surgery or femoral endarterectomy. The subjects are instructed to shower with the sodium hypochlorite body wash daily, or as modified by the physician, for 5 of the 7 days leading to their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female greater than the age of 18 years.
2. Subject is willing and able to give written informed consent and to comply with the requirements of the study.
3. Subject has 5 or more days of time prior to elective surgery scheduled to sign consent and begin washing parameters.
4. Subject is capable of taking a shower and lathering their entire body, or is able to be helped by a caregiver to shower each day with lather on their entire body for 5 out of 7 days immediately prior to elective surgery. (Modifications for bath usage can be made by the physician if the result of the product being left on the skin of the entire body for the time commitment is maintained, and if the body can be rinsed with poured water. Bed bath is not considered an allowable modification.)

Exclusion Criteria:

* 1) Subject is on antibiotics prior to surgery.

  2) Subject is unable to maintain washing regimen for the full study term.

  3) Subject is unable to follow pre-surgery cleansing instructions for 5 of the 7 days immediately prior to surgery. (Bed bath is not considered a cleansing day.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in percentage | 5 week per subject
  Fewer infected patients than in the retrospective data

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Hohmann, MD, Principal Investigator — Texas Vascular Associates
Locations (1):
- Texas Vascular Associates, PA, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No